CLINICAL TRIAL: NCT04919499
Title: A First in Human Trial to Study Safety and Tolerability of Single Rising Intravitreal Doses (oPen Label, Non-randomized, Uncontrolled) and in Addition the Early Biological Response of mulTiple Intravitreal Doses (Double-masked, RandomIzed, Sham-controlleD) of BI 765128 in Panretinal photocoaGulation (PRP) Treated Diabetic rEtinopathy (DR) Patients With Diabetic Macular Ischemia (DMI) - the PARTRIDGE Study
Brief Title: A Study of BI 765128 in Patients With an Eye Condition Called Diabetic Macular Ischemia Who Have Received Laser Treatment
Acronym: PARTRIDGE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1451-0001; 2020-005425-87 (EudraCT Number)
Record Dates: First submitted 2021-06-08; First posted 2021-06-09 (Actual); Results first posted 2024-08-27 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Description to masking:
  In Part A no masking will be performed. In Part B participant and investigator will be masked.
  Description to randomisation:
  In Part A no randomisation will be performed. In Part B randomisation will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single rising dose part: low-dose BI 765128 (Experimental): Diabetic retinopathy (DR) patients with Diabetic Macular Ischemia (DMI) previously treated with panretinal photocoagulation (PRP) received one single intravitreal injection of low-dose BI 765128.
  Interventions: Drug: BI 765128
- Single rising dose part: medium-dose BI 765128 (Experimental): Diabetic retinopathy (DR) patients with Diabetic Macular Ischemia (DMI) previously treated with panretinal photocoagulation (PRP) received one single intravitreal injection of medium-dose BI 765128.
  Interventions: Drug: BI 765128
- Single rising dose part: high-dose BI 765128 (Experimental): Diabetic retinopathy (DR) patients with Diabetic Macular Ischemia (DMI) previously treated with panretinal photocoagulation (PRP) received one single intravitreal injection of high-dose BI 765128.
  Interventions: Drug: BI 765128
- Multiple dose part: high-dose BI 765128 (Experimental): Diabetic retinopathy (DR) patients with Diabetic Macular Ischemia (DMI) previously treated with panretinal photocoagulation (PRP) received 3 single intravitreal injection of high-dose BI 765128 at week 1, 4 and 8.
  Interventions: Drug: BI 765128
- Multiple dose part: Sham (Sham Comparator): Diabetic retinopathy (DR) patients with Diabetic Macular Ischemia (DMI) previously treated with panretinal photocoagulation (PRP) received 3 single intravitreal sham injection at week 1, 4 and 8.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Drug: BI 765128 — BI 765128
  Arms: Multiple dose part: high-dose BI 765128; Single rising dose part: high-dose BI 765128; Single rising dose part: low-dose BI 765128; Single rising dose part: medium-dose BI 765128
Other: Sham comparator — Sham comparator
  Arms: Multiple dose part: Sham

SUMMARY:
This study is open to adults with diabetic macular ischemia who have received laser treatment. The main purpose of this study is to find out whether people with diabetic macular ischemia can tolerate a medicine called BI 765128.

In this study, BI 765128 is given to people for the first time.

The study has 2 parts. Part A tests 3 doses of BI 765128. Participants get either a low, medium or high dose of BI 765128 as a single injection into the eye. If participants tolerate it well, the highest dose will be used in part B.

In part B, participants are put into 2 groups randomly, which means by chance. 1 group gets BI 765128 as injection into the eye. The other group gets sham injections. A sham injection means that it is not a real injection and contains no medicine. Participants cannot tell whether they get the real injection or a sham injection. In this part, participants receive study treatment once every month for 3 months.

Participants in part A are in the study for about 4 months and visit the study site about 8 times.

Participants in part B are in the study for about 5 months and visit the study site about 7 times.

The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Panretinal photocoagulation-treated diabetic retinopathy (DR) patients with either no or inactive retinal neovascularization per investigator judgement in the study eye
* Male or female subjects of age ≥ 18 years
* Evidence of diabetic macular ischemia (DMI) per investigator´s judgement, defined as any degree of disruption of retinal vascularity in optical coherent tomography angiography (OCTA)
* Glycosylated Hemoglobin, Type A1C (HbA1c) of ≤ 12.0%
* Best-corrected visual acuity (VA) ≤75 letters (20/32) in the study eye
* Best corrected visual acuity (VA) in the non-study eye must be equal to or better than best corrected VA in the study eye. If both eyes are eligible and have identical best corrected VA the investigator may select the study eye.
* Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use two methods of contraception with at least one of them being a highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Part B:

* Panretinal photocoagulation-treated diabetic retinopathy (DR) patients with either no or inactive retinal neovascularization per investigator judgement
* Male or female subjects of age ≥ 18 years
* Presence of significant diabetic macular ischemia (DMI): Large foveal avascular zone (FAZ) defined as those with ≥0.5mm2 area present on optical coherent tomography angiography (OCTA). If FAZ is <0.5mm2 then an enlarged peri-foveal inter-capillary space in at least 1 quadrant will be sufficient.
* Glycosylated Hemoglobin, Type A1C (HbA1c) of ≤ 12.0%
* Best-corrected visual acuity (VA) ≤85 letters (20/20) in the study eye
* If both eyes are eligible, the investigator may select either eye to be the study eye.
* Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use two methods of contraception with at least one of them being a highly effective method of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

Part A:

* Subjects receiving intravitreal (IVT) injections for active Diabetic Macular Edema (DME) (anti-vascular endothelial growth factor (VEGF), steroids) and macular laser in the previous 3 months to screening in the study eye
* Subjects receiving anti-VEGF IVT injections for active diabetic retinopathy (DR) in the previous 3 months to screening in the study eye
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoxamine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol)
* Additional progressive eye disease in the study eye that could compromise best corrected visual acuity (VA) (best corrected visual acuity (BCVA)), uncontrolled glaucoma (intra-ocular pressure (IOP)>24), history of high myopia > 8 diopters in the study eye. Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with spectral domain optical coherence tomography (SD-OCT) and optical coherent tomography angiography (OCTA).
* Any intraocular surgery in the study eye within 3 months prior to screening
* Glaucoma tube shunts
* Aphakia or total absence of the posterior capsule. Yttrium aluminum garnet (YAG) laser capsulotomy permitted, if completed more than 3 months prior to screening, in the study eye
* Subjects not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator´s opinion, makes the subject an unreliable trial subject) Further exclusion criteria apply

Part B:

* Diabetic Macular Edema (DME), defined as a Central Subfield Thickness (CST) ≥ 305μm for men and ≥ 290 μm for women (Optovue Angiovue) in the study eye
* Subjects receiving intravitreal (IVT) injections for active DME (anti-vascular endothelial growth factor (VEGF), steroids) and macular laser in the previous 3 months to screening in the study eye
* Subjects receiving anti-VEGF intravitreal IVT injections for active Diabetic Retinopathy (DR) in the previous 3 months to screening in the study eye
* Heavily lasered macula in the study eye per investigator judgement
* History of vitrectomy in the study eye
* Epiretinal membrane with extended foveal contour distortion in the study eye
* Current or planned use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoxamine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, nicotinic acid, and ethambutol)
* Additional eye disease in the study eye that could compromise best corrected VA (BCVA). Significant visual field loss, uncontrolled glaucoma (IOP>24), clinically significant diabetic maculopathy, history of ischemic optic neuropathy or retinal vascular occlusion, symptomatic vitreomacular traction, or genetic disorders such as retinitis pigmentosa; history of high myopia > 8 diopters in the study eye. Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation with SD-OCT and OCTA Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (11):
  - California Retina Consultants, Bakersfield, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Cumberland Valley Retina Consultants, PC., Hagerstown, Maryland
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Austin Research Center for Retina, PLLC, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
- Australia (2):
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
- Riga East University Hospital, Riga, Latvia
- Leids Universitair Medisch Centrum (LUMC), Leiden, Netherlands
- Spain (4):
  - Hospital Dos de Maig, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (6):
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital, London
  - Central Middlesex Hospital, London
  - Oxford Eye Hospital, Oxford
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a trial consisting of a non-randomised, uncontrolled, open label single rising dose part (Part A) and a randomised, sham controlled, double-masked multiple doses part (Part B).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. One eye was selected, according to inclusion /exclusion criteria, as the study eye to be treated.
Period: Overall Study
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128 | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Started | 3 | 3 | 6 | 11 | 23
Treated | 3 | 3 | 6 | 10 | 23
Completed | 3 | 3 | 6 | 10 | 21
Not Completed | 0 | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Not treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) - all subjects who were treated with at least one dose of study drug in the single rising dose part and all subjects who were randomized and treated with at least one dose of study drug (either treatment with BI 765128 or Sham) in the multiple dose part.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128 | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 10 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.7 (9.0) | 50.7 (14.4) | 63.8 (6.7) | 52.0 (15.5) | 57.7 (12.4) | 57.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 4 | 9 | 18
  Male | 3 | 2 | 2 | 6 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 4 | 7
  Not Hispanic or Latino | 3 | 3 | 5 | 8 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 3
  White | 3 | 3 | 4 | 9 | 21 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Single Rising Dose Part - Number of Subjects With Ocular Dose Limiting Events (DLEs) From Drug Administration Until Day 8 (7 Days After Treatment)
Description: Dose limiting events were defined in the clinical trial protocol as any of the following occurrences in the eye being studied during the evaluation period:
  * development of sterile endophthalmitis and/or sterile inflammation of the vitreous of 3+ (out of 0, 0.5+,1+,2+,3+ and 4+, where 0 is clear vitreous and 4+ is an obscured vitreous) according to the NEI (National Eye Institute) Grading of vitreous haze, and anterior chamber cells of 3+ (out of 0, 0.5+,1+,2+,3+ and 4+, where 0 is no inflammation and 4+ is severe inflammation) according to the Standardization of Uveitis Nomenclature (SUN) working group (WG) grading scheme for 5 or more days;
  * visual loss of more than 15 letters at any given time-point; persistent intra-ocular pressure over 30 mmHg for 3 days;
  * and signs of vascular occlusion in a first (the main branch) or second degree (the vessel after the first bifurcation of the main branch) retinal vessel.
Time Frame: From initial drug administration (day 1) until day 8.
Population: Treated set (TS) - single rising dose part: all subjects who were treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Multiple Dose Part - Number of Subjects With Drug Related Adverse Events (AEs) From Drug Administration Until End of Study (EOS)
Description: Number of subjects with adverse events assessed as drug related by the investigator from first drug administration to end of the multiple dose part of the study.
Time Frame: From first drug administration to end of the multiple dose part of the study, i.e., up to day 141±7.
Population: Treated set (TS) - multiple dose part: all subjects who were randomized and treated with at least one dose of study drug (either treatment with BI 765128 or Sham).
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 10 | 23
Participants | 0 | 1

3. Secondary Outcome: Single Rising Dose Part - Number of Subjects With Drug Related Adverse Events (AEs) at End of Study (EOS)
Description: Number of subjects with adverse events assessed as drug related by the investigator from first drug administration to end of the single rising dose part of the study.
Time Frame: From first drug administration to end of the single rising dose part of the study, i.e., up to day 99±7.
Population: Treated set (TS) - single rising dose part: all subjects who were treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: Single Rising Dose Part - Number of Subjects With Any Ocular Adverse Events (AEs) (Eye Disorders) at End of Study (EOS)
Description: Number of subjects with any ocular adverse events at the end of the single rising dose part of the study.
Time Frame: From first drug administration to end of the single rising dose part of the study, i.e., up to day 99±7.
Population: Treated set (TS) - single rising dose part: all subjects who were treated with at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 1 | 1

5. Secondary Outcome: Multiple Dose Part - Change From Baseline of the Size of the Foveal Avascular Zone (FAZ) in Optical Coherence Tomography Angiography (OCTA) at Visit 5
Description: This outcome measured the change in size of the foveal avascular zone (FAZ) from baseline to visit 5 of the multiple dose part of the trial by optical coherence tomography angiography (OCTA). Results were calculated as [Visit 5] -[Baseline].
  A mixed model with repeated measurements (MMRM) was used for the analysis with fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.
Time Frame: MMRM included measurements at baseline, day 29±3, day 57±3, day 85±7, day 113±7 and day 141±7. Change from baseline values at day 85±7 (visit 5) is reported.
Population: Treated set (TS) - multiple dose part: all subjects who were randomized and treated with at least one dose of study drug (either treatment with BI 765128 or Sham). Only subjects with baseline and at least one on-treatment post baseline value were included in the analysis. Only subjects with measurements with scan quality index 6 or higher were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: millimeter^2
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 7 | 12
millimeter^2 | 0.0075 (0.0302) | -0.0177 (0.0225)
Statistical Analysis 1: Comparison: Multiple Dose Part: Sham vs Multiple Dose Part: High-dose BI 765128; Test type: Other — A mixed model with repeated measurements (MMRM) was used for the analysis with fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors; Adjusted mean difference = -0.0252, 95% CI 2-sided [-0.1048 to 0.0545], Standard Error of Mean 0.0376 — Calculated as [high-dose BI 765128] - [Sham]

6. Secondary Outcome: Multiple Dose Part - Change From Baseline of the Size of the Foveal Avascular Zone (FAZ) in Optical Coherence Tomography Angiography (OCTA) at Visit 6
Description: This outcome measured the change in size of the foveal avascular zone (FAZ) from baseline to visit 6 of the multiple dose part of the trial by optical coherence tomography angiography (OCTA). Results were calculated as [Visit 6] - [Baseline].
  A mixed model with repeated measurements (MMRM) was used for the analysis with fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.
Time Frame: MMRM included measurements at baseline, day 29±3, day 57±3, day 85±7, day 113±7 and day 141±7. Change from baseline values at day 113±7 (visit 6) is reported.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimeter^2
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 8 | 12
millimeter^2 | -0.0020 (0.0189) | -0.0121 (0.0142)
Statistical Analysis 1: Comparison: Multiple Dose Part: Sham vs Multiple Dose Part: High-dose BI 765128; Test type: Other — [test comment as in outcome 5, analysis 1]; Adjusted mean difference = -0.0101, 95% CI 2-sided [-0.0625 to 0.0422], Standard Error of Mean 0.0236 — Calculated as [high-dose BI 765128] - [Sham]

7. Secondary Outcome: Multiple Dose Part - Change From Baseline of the Size of the Foveal Avascular Zone (FAZ) in Optical Coherence Tomography Angiography (OCTA) at Visit 7
Description: This outcome measured the change in size of the foveal avascular zone (FAZ) from baseline to visit 7 of the multiple dose part of the trial by optical coherence tomography angiography (OCTA). Results were calculated as [Visit 7] - [Baseline].
  A mixed model with repeated measurements (MMRM) was used for the analysis with fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.
Time Frame: MMRM included measurements at baseline, day 29±3, day 57±3, day 85±7, day 113±7 and day 141±7. Change from baseline values at day 141±7 (visit 7) is reported.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimeter^2
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 8 | 11
millimeter^2 | -0.0087 (0.0135) | -0.0071 (0.0120)
Statistical Analysis 1: Comparison: Multiple Dose Part: Sham vs Multiple Dose Part: High-dose BI 765128; Test type: Other — [test comment as in outcome 5, analysis 1]; Adjusted mean difference = 0.0016, 95% CI 2-sided [-0.0504 to 0.0536], Standard Error of Mean 0.0181 — Calculated as [high-dose BI 765128] - [Sham]

8. Secondary Outcome: Multiple Dose Part - Change From Baseline of Best Corrected Visual Acuity (BCVA) at Visit 7
Description: This outcome measured the absolute change in best corrected visual acuity (BCVA) from baseline to visit 7 of the multiple dose part of the trial. The BCVA was measured using the early treatment diabetic retinopathy study (ETDRS) visual acuity chart. The BCVA score was the number of letters read correctly by the patient. Results were calculated as [Visit 7] - [Baseline] and were rounded to one decimal place.
  A mixed model with repeated measurements (MMRM) was used for the analysis with fixed, categorical effects of treatment at each visit and the fixed continuous effects of baseline at each visit. Visit was treated as the repeated measure with an unstructured covariance structure used to model the within-patient measurements. The Kenward-Roger approximation was used to estimate denominator degrees of freedom and adjust standard errors.
Time Frame: as for outcome 7
Population: Treated set (TS) - multiple dose part: all subjects who were randomized and treated with at least one dose of study drug (either treatment with BI 765128 or Sham). Only subjects with baseline and at least one on-treatment post baseline value were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Number of letters
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 10 | 20
Number of letters | 1.1 (1.9) | 1.3 (1.3)
Statistical Analysis 1: Comparison: Multiple Dose Part: Sham vs Multiple Dose Part: High-dose BI 765128; Test type: Other — [test comment as in outcome 5, analysis 1]; Adjusted mean difference = 0.1, 95% CI 2-sided [-4.7 to 5.0], Standard Error of Mean 2.4 — Calculated as [high-dose BI 765128] - [Sham] Results were rounded to one decimal place

9. Secondary Outcome: Multiple Dose Part - Number of Subjects With Any Ocular Adverse Events (AEs) (Eye Disorders) From Drug Administration Until End of Study (EOS)
Description: Number of subjects with any ocular adverse events at the end of the multiple dose part of the study.
Time Frame: From first drug administration to end of the multiple dose part of the study, i.e., up to day 141±7.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
Number analyzed (Participants) | 10 | 23
Participants | 3 | 9

ADVERSE EVENTS:
Time Frame: Single rising dose part: From first drug administration to end of study, i.e., up to day 99±7. Multiple dose part: From first drug administration to end of study, i.e., up to day 141±7.
Description: Treated set (TS) - all subjects who were treated with at least one dose of study drug in the single rising dose part and all subjects who were randomized and treated with at least one dose of study drug (either treatment with BI 765128 or Sham) in the multiple dose part.
Arm/Group | Single Rising Dose Part: Low-dose BI 765128 | Single Rising Dose Part: Medium-dose BI 765128 | Single Rising Dose Part: High-dose BI 765128 | Multiple Dose Part: Sham | Multiple Dose Part: High-dose BI 765128
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/10 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/6 | 2/10 | 3/23
Other Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 3/6 | 5/10 | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Rising Dose Part: Low-dose BI 765128 (N=3) | Single Rising Dose Part: Medium-dose BI 765128 (N=3) | Single Rising Dose Part: High-dose BI 765128 (N=6) | Multiple Dose Part: Sham (N=10) | Multiple Dose Part: High-dose BI 765128 (N=23)
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Rising Dose Part: Low-dose BI 765128 (N=3) | Single Rising Dose Part: Medium-dose BI 765128 (N=3) | Single Rising Dose Part: High-dose BI 765128 (N=6) | Multiple Dose Part: Sham (N=10) | Multiple Dose Part: High-dose BI 765128 (N=23)
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT04919499/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT04919499/SAP_001.pdf